CLINICAL TRIAL: NCT00159666
Title: A Double-Blind Randomized Placebo-Controlled Trial of the Time to Onset of Pain Relief in Subjects With Post Therapeutic Neuralgia (PHN) Treated With Pregabalin (150 - 600 Mg/Day Flexible Optimized Dose or 300 Mg/Day Fixed Dose) or Placebo
Brief Title: Study of Pregabalin Therapy for Pain Relief in Subjects With Post-Herpetic Neuralgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081004
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2006-11

CONDITIONS: Post-Herpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin

INTERVENTIONS:
Drug: pregabalin

SUMMARY:
The purpose of this study is to measure how rapidly pregabalin treatment can relieve pain in patients with post-herpetic neuralgia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PHN with pain present for at least three months after the healing of a Herpes Zoster skin lesion.
* Subjects must have completed the Daily Pain Rating Scale in the electronic diary at least 4 times during screening and have an average daily pain rating score of greater than or equl to 4 during the 7 +/- 3 days prior to randomization (Visit 2).

Exclusion Criteria:

* History of neurolytic or neurosurgical therapy for PHN.
* Presence of any severe pain associated with conditions other than PHN that may confound the assessment or self-evaluation of the pain due to PHN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255
Dates: Start 2004-10; Study Completion 2006-06

PRIMARY OUTCOMES:
Onset meaningful pain reduction

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (14):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Oak Brook, Illinois
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
- Germany (10):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bochum
  - Pfizer Investigational Site, Düsseldorf
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Göppingen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hattingen
  - Pfizer Investigational Site, Jena
  - Pfizer Investigational Site, Nuremberg
  - Pfizer Investigational Site, Wiesbaden
- Italy (4):
  - Pfizer Investigational Site, L’Aquila
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pisa
  - Pfizer Investigational Site, Roma
- Spain (6):
  - Pfizer Investigational Site, Leganés, Madrid
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Granada
  - Pfizer Investigational Site, Salamanca
  - Pfizer Investigational Site, Seville
  - Pfizer Investigational Site, Valencia
- United Kingdom (6):
  - Pfizer Investigational Site, Middlesbrough, Cleveland
  - Pfizer Investigational Site, Addlestone, Surrey
  - Pfizer Investigational Site, Chicester, Sussex
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Oldham, Lancashire
  - Pfizer Investigational Site, Portsmouth

REFERENCES:
- [Derived] Schug SA, Parsons B, Almas M, Whalen E. Effect of Concomitant Pain Medications on Response to Pregabalin in Patients with Postherpetic Neuralgia or Spinal Cord Injury-Related Neuropathic Pain. Pain Physician. 2017 Jan-Feb;20(1):E53-E63. PMID 28072797
- [Derived] Markman JD, Jensen TS, Semel D, Li C, Parsons B, Behar R, Sadosky AB. Effects of Pregabalin in Patients with Neuropathic Pain Previously Treated with Gabapentin: A Pooled Analysis of Parallel-Group, Randomized, Placebo-controlled Clinical Trials. Pain Pract. 2017 Jul;17(6):718-728. doi: 10.1111/papr.12516. Epub 2016 Dec 1. PMID 27611736
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081004&StudyName=Study+of+Pregabalin+Therapy+for+Pain+Relief+in+Subjects+with+Post%2DHerpetic+Neuralgia